CLINICAL TRIAL: NCT04968340
Title: External Pop Out Caesarean Section Versus Conventional Method for Fetal Head Extraction in Repeated Caesarean Section, a Randomized Controlled Trial.
Brief Title: External Pop Out cs vs Conventional Method for Fetal Head Extraction in Repeatedcaesarean Section.
Acronym: EPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Azhar Samir Aboelfadl, director, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPO technique
Record Dates: First submitted 2021-06-16; First posted 2021-07-20 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: EPO Teqnique in Fetal Head Extraction

STUDY DESIGN:
Intervention Model Description: Support of the lower uterine segment and bladder without introduction of the obstetrician hand in the uterine incision so as not to occupy more space ; this help rotation of the foetal head facilitating head delivery, protecting LUS incision from extension.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- • Group 1(conventional c s) (Other): this arm will be exposed to the conventional method of cesserian section which entail introduction of the operator hand below the fetal head during its extraction
- • Group2(EPO technique) (Other): this group will be exposed to external pop out teqnique which entails support of lower uterine segment without introduction of the obstetrician hand into uterine incision

INTERVENTIONS:
Procedure: conventional cs — after opening the lower uterine segment, introduction of the surgeon fingers inside the uterus below the fetal head during its extraction
Procedure: external pop out teqnique — support of lower uterine segment from outside without introduction of the surgeon fingers inside the uterus, guiding the fetal head to pop out from the uterine incision

SUMMARY:
To establish feasibility and safety of the use of external pop out as a novel technique for foetal head delivery during c s, the effect of application of this method on a previously scarred uterus will be studied as a better way regarding preservation of the integrity of the lower uterine segment, operative time, time needed for head delivery, incision extension, blood loss, incidence of bladder injury.

DETAILED DESCRIPTION:
Caesarean delivery (cs) is the most common major surgical procedure performed with over 1,2million performed per year . The increase in caesarean section rates seems uncontrollable with no signs that it is slowing down .

A great concern of caesarean delivery complications is incision extension , un intended extensions of uterine incision frequently occurs at the time of caesarean delivery with estimated incidence of 4-8% .

Some measures are taken to guard against incision extension as expansion of uterine incision in cephalocaudal direction which is associated with lower risk of un intended extension Head extraction during caesarean section is one of the most critical steps during caesarean section and one of the major contributors to un intended uterine incision extension . Delivery of the foetal head should be within 3minutes from opening the uterine incision.

Difficult extraction causes different hazards as foetal respiratory distress syndrome , incision extension, bleeding.

The original technique of foetal head extraction entails introduction of obstetrician hands or other instruments into lower uterine segment (LUS) .

Criticizing the standard:

Insertion of obstetrician hand inside the uterine incision will occupy more space and this will increase possibility of incision extension and puts the LUS at risk of damage and increased blood loss, increased operative time , Interfere with head rotation &repositioning of the head may happen during head delivery leading to difficult extraction.

Inadequate opening will add more pressure on uterine incision increasing possibility of extension.

In cases of repeated c s , lower uterine segment is thin, adherent to the urinary bladder this makes the conventional method of head extraction unreliable causing more bleeding, extension, bladder injury, more operative time, postoperative adhesions.

The rational of EPO technique:

Support of the lower uterine segment and bladder without introduction of the obstetrician hand in the uterine incision so as not to occupy more space ; this help rotation of the foetal head facilitating head delivery, protecting LUS incision from extension.

Preoperative sonographic assessment of the lower uterine segment thickness will be done within two weeks of delivery using transabdominal us with critical cut off value of 2.5 mm which is associated with dehiscent scar according to ROC curve.

ELIGIBILITY:
Inclusion Criteria:

* Cases with repeated c s.
* Elective c s.
* Singleton pregnancy.
* Full term pregnancy.

  -BMI below30
* Cephalic presentation.
* Women who accepted to participate in the study.
* Placenta away from the lower segment

Exclusion Criteria:

* Fibroid uterus.
* Infection as chorioamnionitis.
* Maternal comorbidities.
* Uterine anomalies.
* Major Foetal congenital anomalies.
* Placenta previa.

Placental separation.

Dehiscent LUS scar as assessed by us with cut off value 2.5mm.

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women full term with repeated cs
Enrollment: 600 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-07-24 (Actual); Study Completion 2022-08-28 (Actual)

PRIMARY OUTCOMES:
Rate of uterine incision extension or LUS injury | through the study completion average one year
  The percentage of participants who developed uterine incision extension or lower uterine segment injury in both groups of study.

SECONDARY OUTCOMES:
The degree of severity of incision extension or injury | through the study completion average one year
  measuring the extension or injury in cm or associated bladder or uterine artery injury
Amount of intraoperative blood loss | through the study completion average one year
  Number of towels used in the hemostasis during repair of the incison or an extension/injury
Total operative time and uterotomy to head delivery time | through the study completion average one year
  Total time of whole surgery and the time from uterine incision and head delivery in minutes
Post operative hemoglobin level | 24 hours postoperative in each participant through the study completion average one year
  Estimation of HB level (gm/dl) after 24 hours postoperative
Need for blood transfusion | Intraoperative or postoperative before discharge from the hospital
  excessive intraoperative blood loss or affected vitals of the patient
Hospital stay | Through the study completion average one year
  Postoperative hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Hisham abou taleb, professor, Study Director — Assiut University
Locations (1):
- Faculty of Medicine, Obstetrics and Gynecology department, Assiut University, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The anonymized participants data and study protocols can be shared after publication when reasonably requested .These data will be available also for other qualified researchers after publication as an accessory data at the site of publishing journal.
Supporting Information: Study Protocol, SAP
Time Frame: After publication

REFERENCES:
- [Background] Berghella V, Baxter JK, Chauhan SP. Evidence-based surgery for cesarean delivery. Am J Obstet Gynecol. 2005 Nov;193(5):1607-17. doi: 10.1016/j.ajog.2005.03.063. PMID 16260200
- [Background] Fioretti BT, Reiter M, Betran AP, Torloni MR. Googling caesarean section: a survey on the quality of the information available on the Internet. BJOG. 2015 Apr;122(5):731-9. doi: 10.1111/1471-0528.13081. Epub 2014 Sep 11. PMID 25209160